CLINICAL TRIAL: NCT03471065
Title: A Prospective, Single-arm, Multicenter Study of the SAPIEN 3 Ultra System in Intermediate Risk Patients With Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: The SAPIEN 3 Ultra System in Intermediate Risk Patients With Symptomatic, Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-03
Record Dates: First submitted 2018-03-05; First posted 2018-03-20 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter; Transcatheter Valve Replacement; SAPIEN 3 Ultra
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: SAPIEN 3 Ultra System
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental)
  Interventions: Device: SAPIEN 3 Ultra Delivery System with the SAPIEN 3 Ultra THV

INTERVENTIONS:
Device: SAPIEN 3 Ultra Delivery System with the SAPIEN 3 Ultra THV — Patients will be implanted with the SAPIEN 3 Ultra THV (20, 23 and 26 mm) or SAPIEN 3 THV (29 mm) using the SAPIEN 3 Ultra Delivery System.

SUMMARY:
This study will confirm the procedural safety and performance of the SAPIEN 3 Ultra System in subjects with severe, calcific AS who are at intermediate operative risk for standard aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Severe, calcific aortic stenosis meeting the following transthoracic echocardiogram criteria:

   * Aortic valve area ≤ 1.0 cm2 OR aortic valve area index ≤ 0.6 cm2/m2
   * Jet velocity ≥ 4.0 m/s OR mean gradient ≥ 40 mmHg
2. New York Heart Association functional class ≥ II
3. Judged by the Heart Team to be at intermediate risk for open surgical therapy
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Native aortic annulus size unsuitable for available THV sizes on 3D imaging analysis
2. Aortic valve is unicuspid, bicuspid or non-calcified
3. Pre-existing mechanical or bioprosthetic valve in any position.
4. Severe aortic regurgitation (> 3+)
5. Severe mitral regurgitation (> 3+) or ≥ moderate stenosis
6. Ventricular dysfunction with left ventricular ejection fraction < 30%
7. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
8. Evidence of an acute myocardial infarction ≤ 30 days before the valve implant procedure
9. Subjects with planned concomitant ablation for atrial fibrillation
10. Hypertrophic cardiomyopathy with obstruction
11. Coronary anatomy that increases the risk of coronary artery obstruction post-TAVR
12. Complex coronary artery disease:

    1. Unprotected left main coronary artery
    2. SYNTAX score > 32
    3. Heart Team assessment that optimal revascularization cannot be performed
13. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath
14. Significant abdominal or thoracic aortic disease that would preclude safe passage of the delivery system
15. Active bacterial endocarditis within 180 days of the valve implant procedure
16. Stroke or transient ischemic attack within 90 days of the valve implant procedure
17. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of the valve implant procedure
18. Severe lung disease (Forced Ejection Volume 1 < 50% predicted) or currently on home oxygen
19. Severe pulmonary hypertension
20. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of the valve implant procedure
21. History of cirrhosis or any active liver disease
22. Renal insufficiency and/or renal replacement therapy at the time of screening
23. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy or hypercoagulable states
24. Inability to tolerate or condition precluding treatment with antithrombotic therapy during or after the valve implant procedure
25. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
26. Significant frailty as determined by the Heart Team
27. Subject refuses blood products
28. Body mass index > 50 kg/m2
29. Estimated life expectancy < 24 months
30. Positive urine or serum pregnancy test in female subjects of childbearing potential
31. Currently participating in an investigational drug or another device study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Webb, MD, Principal Investigator — St. Paul's Hospital; Bernard Prendergast, Prof, Principal Investigator — St. Thomas Hospital
Locations (6):
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
- United Kingdom (2):
  - Kings Hospital, London
  - St. Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.5 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Society of Thoracic Surgeons (STS) Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk of operative mortality.
  units on a scale | 3.6 (1.29)
New York Heart Association (NYHA) Class Grouped [Count of Participants; unit: Participants] — New York Heart Association (NYHA) functional classification of heart failure is based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
  Participants
    Class I/II | 56
    Class III/IV | 44

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: The number of patients with procedural success, defined as freedom from all of the following at exit from the procedure room:
  * Mortality
  * Conversion to surgery
  * Moderate or severe paravalvular regurgitation
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 100
Participants | 100

2. Secondary Outcome: Major Vascular Complications
Description: Number of patients with major vascular complications
Time Frame: Discharge, expected to be within 1-5 days post-procedure]
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 100
Participants | 2

3. Secondary Outcome: Valve Migration or Embolization
Description: Number of patients with valve migration or embolization
Time Frame: Discharge, expected to be within 1-5 days post-procedure]
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 100
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Transcatheter Aortic Valve Replacement (TAVR)
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 28/100
Other Adverse Events (participants affected / at risk) | 14/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Aortic Valve Replacement (TAVR) (N=100)
Atrioventricular block complete (Cardiac disorders) | 7 (7)
Atrioventricular block first degree (Cardiac disorders) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bundle branch block bilateral (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 3 (3)
Sinus arrest (Cardiac disorders) | 1 (1)
Ventricular asystole (Cardiac disorders) | 1 (1)
Prosthetic cardiac valve stenosis (General disorders) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 2 (2)
Femoral artery perforation (Vascular disorders) | 1 (1)
Iliac artery perforation (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Aortic Valve Replacement (TAVR) (N=100)
Bundle branch block left (Cardiac disorders) | 8 (8)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT03471065/Prot_SAP_000.pdf